CLINICAL TRIAL: NCT01163123
Title: Seroepidemiology of Japanese Encephalitis Virus Infection in Hualien, Taiwan
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Mennonite Christian Hospital (Other)
Responsible Party: Sheng-Hsuan Chen, Mennonite Christian Hospital
Other Study IDs: D9902
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Last update posted 2010-07-16 (Estimated); Status verified 2010-07

CONDITIONS: Japanese Encephalitis
Keywords: Subclinical infection of Japanese encephalitis virus
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The sera from volunteer was collected to detect IgG, IgM and anti-NS1 antibody against Japanese encephalitis virus
Oversight: Data Monitoring Committee: No

SUMMARY:
Japanese encephalitis (JE) is one of important zoonotic infectious diseases in Taiwan. JE caused by Japanese encephalitis virus (JEV) which transmitted by Culex tritaeniorhynchus and used swine as amplifying host. Infections leading to overt encephalitis are estimated to be 1 in 1000 cases. Among JE confirmed cases, approximately 25 percent of cases die and 50 percent of the survivals develop permanent neurologic and/or psychiatric sequelae. JEV circulated in Taiwan are belonged to genotype III and the vaccine strain selected from same genotype. Genotype I JEV was first detected in northern Taiwan in 2008 by CDC, and the same genotype JEV were detected in mosquito collected in central Taiwan by our group. In order to study the genotypic shift of JEV in Taiwan areas, and the effects of the replacement of genotype on vaccine, we will conduct the JEV seroepidemiology in Hualien county which was the highest incidence of JEV in Taiwan. The aims of this study were: (1) study the circulating of genotype I JEV in Hualien county; (2) determine the virulence of genotype I JEV in human; (3) differential diagnosis of JEV genotype I or III infection among confirmed cases; (4) measure the cross neutralizing activity, after immunized with genotype III JEV vaccine, against genotype I JEV; (5) determine the age-specific seroprevalence of JEV antibody; (6) estimate the annual risk of infection for JEV.

DETAILED DESCRIPTION:
According to CDC Taiwan epidemiology data, Hualien county had 6 confirmed JEV infection patients in 2009 witch was the highest county in Taiwan. Since mass vaccination was arranged since 45 years ago in Taiwan, most of the JEV infection was happened on the elderly, possible due to aging and immune compromised. However, from Mennonite Christian Hospital and CDC records, most of the confirmed JEV patients in Hualien county were aboriginal people. The youngest patient in 2009 is around 30-year-old who lived in the mountain side aboriginal village. Whether aboriginal people are at more risk for JEV infection or Genotype I JEV was appeared in Hualien with more virulent, resistent to vaccine protection is unknown.

In order to understand the risk of JEV infection and environmental (mosquito, swine) surveillance, we had arranged a small cohort study in 2 villages. The 2 villages are located at middle Hualien with direct distance around 20 KM between each other. Both villages had several pig farms and mosquito numbers in summer were very high. Both villages had document JEV infection resident in past 2 years. The first village was near the river ready to entrance the sea (wetlands) and many migrate birds appeared in the summer every year. The residence were mostly Han people. The seconds village was located very closed to the central mountain Taiwan and the residence were almost aboriginal people.

In this year 2010, we plan to do the following research:

1. Collect mosquito in 2 villages since May.2010 with RT-PCT method to identify the JEV genotype
2. Collect sera from swine in 2 villages to identify the JEV genotype
3. Collect sera from 312 residency in 2 villages at May and Sep 2010 to detect sub-clinical infection rate. ( estimated sub-clinical infection rate = 2.5%)
4. Identify the JEV from new diagnosed patient in 2010.

Since virus was hardly detected by RT-PCR or virus isolation from JEV infected patient, the virus identified from mosquito or swine in the nearby may show indirect evidence of the JEV genotype.

After comparing the 2 sera from the same person during the summer in these 2 villages, we can identify:

1. The subclinical infection rate of the JEV (genotype I or III, depends on JEV isolated from mosquito)
2. Whether aboriginal people near the central mountains are at more risk then people near the wetlands.

ELIGIBILITY:
Inclusion Criteria:

1. Living in the specific 2 villages in Hualien county
2. Aged 18-85

Exclusion Criteria:

1. Difficulty to have blood test due to coagulopathy or small blood vessels

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers were recruited from 2 villages in Hualien county Taiwan. There were at least one patient who had confirmed diagnosis of Japanese virus encephalitis in past 2 years. Many pig farms were located in these 2 villages also. The volunteers are either living or working in the villages during 2010 summer. We had blood test for IgM, IgG for Japanese virus encephalitis before and after the summer season to identify possible subclinical infection. At the same time, mosquito were analyzed by RT-PCR periodically to identify possible virus in the community.
Sampling Method: Non-Probability Sample
Enrollment: 312 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Measure the subclinical infection rate in the cohort population during the summer ( May 2010 ~ Sep 2010) | May 2010 - Oct 2010
  We exam 2 sera from volunteer collected seperately on May and October 2010 to estimate the subclinical infection rate. Subclinical infection rate was defined by one of the following
  1. 4 times increased in IgG titer
  2. Appearance of IgM in the second sera
  3. Apperance of Anti-NS1 antibody in the second sera

CONTACTS AND LOCATIONS:
Overall Officials: ChenChang Shih, Study Director